CLINICAL TRIAL: NCT00687869
Title: Participative Rehabilitation Process Management "Stroke in Saxony-Anhalt"
Brief Title: Participative Rehabilitation in Stroke Patients
Acronym: PaReSiS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Forschungsverbund Rehabilitationswissenschaften Sachsen-Anhalt (Unknown); Deutsche Rentenversicherung (Other); Universitätsklinik und Poliklinik für Neurologie (Unknown)
Responsible Party: Principal Investigator, Johann Behrens, Prof. Dr. phil. habil., Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 01GX0711
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; patient care management; patient participation
MeSH Terms: conditions — Stroke; Patient Participation | interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case management (Experimental): Case management with patient-information-notes, telephone hotline, individual counselling using home visits, e-mail and telephone contact, web portal
  Interventions: Behavioral: Case management
- usual care (Active Comparator): Usual stroke aftercare plus patient-information-notes
  Interventions: Behavioral: Case management

INTERVENTIONS:
Behavioral: Case management — Case management with patient-information-notes, telephone hotline, individual counselling using home visits, e-mail and telephone contact, web portal
  Arms: Case management
Behavioral: Case management — Usual stroke aftercare plus patient-information-notes
  Arms: usual care

SUMMARY:
Primary objective of this study is to determine whether a case management of stroke patients after discharge to home or to nursing home results in improving physical and cognitive capacity one year after discharge.

DETAILED DESCRIPTION:
In a randomized trial, the project Participative rehabilitation process management "Stroke in Saxony-Anhalt" (PaReSiS) implements a case management trial, explicitly including all providers in the course of illness, treatment and rehabilitation. To achieve this, patients in the intervention group have the opportunity to choose, specifically and according to their own needs, from the offers of a web portal and a telephone hotline, from individual counselling and info sessions as well as from home visits. Patients in the control group receive patient-information-notes beyond primary care. There will be qualitative interviews with the persons concerned and/or their relatives in both groups in order to validate the instruments.

ELIGIBILITY:
Inclusion Criteria:

* Acute cerebrovascular event (ischemic stroke or intra-cerebral bleeding) with signs and symptoms of an acute stroke according to the diagnosis I61 and I63 of the ICD-10-GM 2008
* Differentiation between ischemic or haemorrhagic stroke by the use of CT or MRT
* Resident in Saxony-Anhalt or Saxony or Thuringia
* Able to understand German language

Exclusion Criteria:

* Reinfarction
* Alcoholism
* Death in acute care
* NIHHS > 25
* Homelessness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2008-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
physical scale of the Stroke Impact Scale 3.0 | before discharge from acute care, four weeks after discharge from the hospital or rehabilitation (in case of referral to a medical rehabilitation) immediately before randomization (baseline assessment), and 12 months after randomization

SECONDARY OUTCOMES:
Health related quality of life, depression, mortality, recurrent stroke and/or TIA/PRIND | before discharge from acute care, four weeks after discharge from the hospital or rehabilitation (in case of referral to a medical rehabilitation) immediately before randomization (baseline assessment), and 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Johann Behrens, Prof. Dr., Principal Investigator — Institute for Health and Nursing Science, Medical faculty, Martin-Luther-University Halle-Wittenberg, Halle (Saale)
Locations (1):
- Institute for Health and Nursing Science, Medical faculty, Martin-Luther-University Halle-Wittenberg, Halle (Saale), Halle, Germany

REFERENCES:
- [Derived] Saal S, Becker C, Lorenz S, Schubert M, Kuss O, Stang A, Muller T, Kraft A, Behrens J. Effect of a stroke support service in Germany: a randomized trial. Top Stroke Rehabil. 2015 Dec;22(6):429-36. doi: 10.1179/1074935714Z.0000000047. Epub 2015 Apr 28. PMID 25920942